CLINICAL TRIAL: NCT02939534
Title: Antigen Presentation and Lymphocyte Response in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Roy Alcalay, Principal Investigator, Columbia University
Other Study IDs: AAAN7912
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; autoimmunity
MeSH Terms: conditions — Parkinson Disease; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD and Controls: 50% of the participants will be healthy controls and 50% will be patients diagnosed with Parkinson's disease

SUMMARY:
The way the immune system responds to certain PD-related proteins in PD donors compared to the way it responds in persons without or fewer PD related proteins is not well studied and this study aims to analyze the autoimmune response in each group. The study involves a one time visit involving brief questionnaires and a blood draw of 30 mL (approximately 2 tablespoons) to be collected.

DETAILED DESCRIPTION:
The role of the immune response in Parkinson's disease (PD) is controversial. Recent studies show that neurons can present MHC-I (major histocompatibility complex - class 1) molecules and therefore may be susceptible to an attack by immune cells. The investigators anticipate that the results of this study will improve our understanding of the mechanisms of immune mediated neuronal degeneration in PD. Initial results suggest that antigens are presented by neuronal MHC-I in PD, and that this could lead to T-cell mediated neuronal death. The most obvious antigen that could be differentially expressed in PD patients and controls would be alpha-synuclein (-syn): -syn oligomers appear in all Lewy bodies and Lewy neurites and are the hallmark of PD changes in the brain. This study will offer the opportunity to further characterize the immune mediated component of PD, and to continue elucidating the biology that underlies antigen presentation and T-cell cytolytic activity.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to advanced PD with classic motor features, and must demonstrate two of the following three: rest tremor, rigidity, or bradykinesia
* Dopaminergic medication benefit (self-reported improvement)
* Age at recruitment: 50 - 90 years
* Age at diagnosis > 47
* PD duration > 3 years
* Willingness to have genotyping and genetic studies as part of laboratory research

Exclusion Criteria:

* Atypical parkinsonism or other neurological disorders
* Recent history of cancer (past 3 years)
* Autoimmune disease (except thyroid disease)
* On chronic immune-modulatory therapy (e.g. SIT (specific immunotherapy), anti-IgE)
* Inability to provide informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinically confirmed Parkinson's disease and age matched controls
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-02; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with T-cell immune response | Day 1-2
  Blood samples from PD patients and controls will be processed. The presence of T cell response against the candidate antigens by patient blood-derived peripheral blood mononuclear cells (PBMC) will be assessed using an enzyme-linked immunosorbent spot (ELISPOT) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Alcalay, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - University of California San Diego School of Medicine, La Jolla, California
  - Shirley Ryan Ability Lab, Chicago, Illinois
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cebrian C, Zucca FA, Mauri P, Steinbeck JA, Studer L, Scherzer CR, Kanter E, Budhu S, Mandelbaum J, Vonsattel JP, Zecca L, Loike JD, Sulzer D. MHC-I expression renders catecholaminergic neurons susceptible to T-cell-mediated degeneration. Nat Commun. 2014 Apr 16;5:3633. doi: 10.1038/ncomms4633. PMID 24736453
- See also: Michael J Fox Foundation ad for study — https://foxtrialfinder.michaeljfox.org/trial/4772/